CLINICAL TRIAL: NCT06945341
Title: International Focus Group-based Discussion on Factors Facilitating an Increased Adoption of Neuromuscular Monitoring.
Brief Title: International Focus Group Discussion on Neuromuscular Monitoring.
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Hugo Carvalho, Research Consultant, AZ Sint-Jan AV
Other Study IDs: FGNMM
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Neuromuscular Blockade; Neuromuscular Block, Residual; Perioperative/Postoperative Complications; Anaesthesiology Devices Associated With Adverse Incidents, Diagnostic and Monitoring Devices
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Postoperative Complications; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1 Central and Eastern Europe: Central and Eastern Europe
  Interventions: Behavioral: Focus-Group discussion
- Group 2 Northern Europe: Northern Europe
  Interventions: Behavioral: Focus-Group discussion
- Group 3 Southern Europe: Southern Europe
  Interventions: Behavioral: Focus-Group discussion
- Group 4 Western Europe: Western Europe
  Interventions: Behavioral: Focus-Group discussion

INTERVENTIONS:
Behavioral: Focus-Group discussion — Focus-Group discussion on factors that could lead to an increase in the adoption of neuromuscular monitoring taking into account different country-specific contexts.

SUMMARY:
Focus-Group based discussion designed to gain more in-depth information on factors that could lead to an increase in the adoption of neuromuscular monitoring taking into account different country-specific contexts.

ELIGIBILITY:
Active EU Anaesthesiologists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active EU Anaesthesiologists
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Thematic analysis | 90 minutes
  Thematic analysis of factors that could lead to an increase in the adoption of neuromuscular monitoring taking into account different country-specific contexts

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint Jan, Bruges, WV, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Focus-Group thematic analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code